CLINICAL TRIAL: NCT02997280
Title: Treatment of Steroid-refractory Acute and Chronic Graft-versus-host Disease With Inhibitor of Janus Kinases
Brief Title: Ruxolitinib for Steroid-refractory GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Collaborators: Ministry of Health, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Ivan S Moiseev, Head of oncology, hematology and transplantation department for adults, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-29-1
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Graft Vs Host Disease
Keywords: acute graft-versus-host disease; chronic graft-versus-host disease; Steroid-refractory GVHD; ruxolitinib; JAK inhibitors
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib treatment (Experimental): Ruxolitinib 10 mg bid for adults and children with body weight > 40 kg, 0.15 mg/kg bid for children with body weight < 40 kg.
  Interventions: Drug: Ruxolitinib Oral Tablet

INTERVENTIONS:
Drug: Ruxolitinib Oral Tablet — Dose reduction criteria for acute GVHD: grade 4 neutropenia or grade 4 thrombocytopenia related to ruxolitinib administration based on the decision of attending physician.
  Dose reduction criteria for chronic GVHD: grade 3 neutropenia, grade 3 thrombocytopenia or anemia requiring transfusion, related to ruxolitinib administration based on the decision of attending physician.
  Reduced dose schedule: 5 mg bid for adults and children with body weight > 40 kg, 0.08 mg/kg bid for children with body weight < 40 kg.
  Treatment discontinuation criteria: complete response; absence of response after 28 days or progressive disease after 7 days for acute GVHD; absence of response after 84 days or progressive disease after 28 days for chronic GVHD; life-threatening complications.

SUMMARY:
Steroid-refractory acute GVHD (srGVHD) is one of the causes of mortality after allogeneic stem cell transplantation, while steroid-refractory chronic GVHD significantly increases morbidity, aggravates quality of life and may also impact survival. Currently there is no standard treatment of srGVHD. One of the most promising agents is Janus kinase (JAK) inhibitor ruxolitinib, which in the retrospective study demonstrated excellent response rate and survival of patients with either acute or chronic srGVHD. This study prospectively evaluates the efficacy of ruxolitinib in srGVHD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of graft-versus-host disease established based on tissue biopsy
* Steroid-refractory acute or chronic graft-versus-host disease according to EBMT/ELN criteria (T. Ruutu et al, 2014)
* Age 1 to 70 years
* Karnofsky index >30%.
* Ability for oral drug intake
* Life expectancy > 1 month
* Signed informed consent

Exclusion Criteria:

* Severe organ dysfunction: AST or ALT >5 upper normal limits (excluding cases related to liver GVHD), creatinine >2 upper normal limits
* Requirement for vasopressor support at the time of enrollment
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Pregnancy
* Somatic or psychiatric disorder making the patient (or legal guardian) unable to sign informed consent

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 84 days
  Partial response for acute GVHD is defined as the improvement of at least one stage in the severity of aGVHD in one organ without deterioration in any other organ. A response had to last for at least 3 weeks. Partial response for chronic GVHD was defined as reduction in GVHD National Institute of Health (NIH) severity score at east for one organ without deterioration in any other organ. A complete response was defined as the absence of any symptoms related to GVHD. Overall response is defined as presence of partial or complete response

SECONDARY OUTCOMES:
6-month overall survival | 6 months
  Time from start of ruxolitinib until death or 6 months, summarized using Kaplan-Meier estimates.
Toxicity based NCI CTC grades | 6 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: nasea, vomiting, anemia, thrombocytopenia, leukopenia, neutropenia, hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), hemorrhagic cystitis (attending physician assessment).
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 6 months
GVHD relapse incidence after complete response | 6 months
  Time from stopping ruxolitinib until recurrence of GVHD or 6 months, summarized using cumulative incidence estimates.
Relapse incidence of underlying hematologic malignancy | 12 months
  Time from starting ruxolitinib until hematologic relapse or 12 months, summarized using cumulative incidence estimates
Quality of life measured by FACT BMT ver. 4 questionnaire in adults | 6 months
Quality of life measured by PedQL Stem Cell transplant module ver.1.0 questionnaire in children | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris V Afanasyev, Prof, Study Director — R.M.Gorbacheva Memorial Institute of Oncology, Hematology and Transplantation, Pavlov First Saint Petersburg State Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeiser R, Burchert A, Lengerke C, Verbeek M, Maas-Bauer K, Metzelder SK, Spoerl S, Ditschkowski M, Ecsedi M, Sockel K, Ayuk F, Ajib S, de Fontbrune FS, Na IK, Penter L, Holtick U, Wolf D, Schuler E, Meyer E, Apostolova P, Bertz H, Marks R, Lubbert M, Wasch R, Scheid C, Stolzel F, Ordemann R, Bug G, Kobbe G, Negrin R, Brune M, Spyridonidis A, Schmitt-Graff A, van der Velden W, Huls G, Mielke S, Grigoleit GU, Kuball J, Flynn R, Ihorst G, Du J, Blazar BR, Arnold R, Kroger N, Passweg J, Halter J, Socie G, Beelen D, Peschel C, Neubauer A, Finke J, Duyster J, von Bubnoff N. Ruxolitinib in corticosteroid-refractory graft-versus-host disease after allogeneic stem cell transplantation: a multicenter survey. Leukemia. 2015 Oct;29(10):2062-8. doi: 10.1038/leu.2015.212. Epub 2015 Jul 31. PMID 26228813